CLINICAL TRIAL: NCT00204113
Title: Integrated Voluntary Control of Unsupported Paraplegic Standing
Brief Title: Control of Unsupported Paraplegic Standing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Glasgow (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GUStandingSCI; UK EPSRC: GR/R79234/01
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-06-13 (Estimated); Status verified 2008-06

CONDITIONS: Spinal Cord Injury; Stroke
Keywords: spinal cord injury; standing; balance; functional electrical stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Stroke

INTERVENTIONS:
Device: Multi-purpose rehabilitation frame
Device: Surface Functional Electrical Stimulation

SUMMARY:
The study will investigate the feasibility of using functional electrical stimulation (FES) of the calf muscles of paraplegic subjects to assist in posture stabilisation during standing. We aim to achieve postural stability by combining controlled FES of the lower-limb muscles with the voluntary motor control skills of the intact upper body.

DETAILED DESCRIPTION:
Aim:

The study will investigate the feasibility of using functional electrical stimulation (FES) of the calf muscles of paraplegic subjects to assist in posture stabilisation during standing. We aim to achieve postural stability by combining controlled FES of the lower-limb muscles with the voluntary motor control skills of the intact upper body.

Background:

In spinal cord injury (SCI), the paralysed muscles generally retain their ability to contract and electrical stimulation can be used in rehabilitation as a therapy. With functional electrical stimulation (FES) the aim is to restore some normal motor functions such as standing, stepping or cycling. A number of studies have investigated the physiological effects and potential therapeutic benefits of lower-limb FES exercise. These studies have shown that the benefits include restoration of muscle bulk and strength, a reduction in the rate of bone demineralisation, improvements in the range of joint motion, and relaxation of spasm. Standing is an important part of rehabilitation therapy for paraplegic patients, and helps to alleviate some of the secondary effects of paralysis.

ELIGIBILITY:
Inclusion Criteria:

* Neurologically intact, healthy individuals individuals with complete spinal cord lesion between T6 and T12

Exclusion Criteria:

* Incomplete SCI

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2002-06

PRIMARY OUTCOMES:
estimates of physical parameters (ie. stiffness, viscosity, inertia)

SECONDARY OUTCOMES:
quality of standing
amount of sway
timing of standing

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J Hunt, BSc, PhD, DSc, Principal Investigator — University of Glasgow
Locations (2):
- United Kingdom (2):
  - University of Glasgow, Glasgow, Lanarkshire
  - Queen Elizabeth National Spinal Injuries Unit, Glasgow, Lanarkshire